CLINICAL TRIAL: NCT01133158
Title: Study Phase II Non-randomized Prospective Open to Assess the Combination of Rituximab, Bendamustine, Mitoxantrone, Dexamethasone (R-BMD) in Patients With Follicular Lymphoma Refractory or Relapsed
Brief Title: R-BMD in Refractory or Relapsed Lymphoma, GELTAMO Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-BMD GELTAMO 08
Record Dates: First submitted 2010-02-11; First posted 2010-05-28 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-02

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Follicular non-Hodgkin's lymphoma relapse refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Bendamustine Hydrochloride; Mitoxantrone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-BMD (Experimental): Rituximab, Bendamustine, Mitoxantrone, Dexamethasone Induction: 6 Rituximab, Bendamustine, Mitoxantrone, Dexamethasone cycles Maintenance: Rituximab every 3 months for 2 years
  Interventions: Drug: Rituximab, Bendamustine, Mitoxantrone, Dexamethasone

INTERVENTIONS:
Drug: Rituximab, Bendamustine, Mitoxantrone, Dexamethasone — Bendamustine: 90 mg/m2/day, days 1 and 2 of each cycle, iv Mitoxantrone: 6 mg/m2/day, day 1 of each cycle, iv Dexamethasone 20 mg / day, days 1 through 5 of each cycle, od Rituximab: 375 mg / m 2 / day, day 1 of each cycle, iv
  Other Names: R-BMD

SUMMARY:
Assess the combination of efficacy of the combination of rituximab, bendamustine, mitoxantrone, dexamethasone in the treatment of patients with Follicular Lymphoma.

DETAILED DESCRIPTION:
Assess the combination of efficacy and safety of the combination of rituximab, bendamustine, mitoxantrone, dexamethasone in the treatment of patients with Follicular Lymphoma who are refractory or in relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years.
2. Patients with follicular lymphoma grade 1, 2 or 3a, CD20 +, histologically confirmed lymph node biopsy or tissue. Be accepted diagnosis in bone marrow if no accessible lymph nodes and whether it has discarded the mantle LLC, and NHL.
3. Follicular lymphoma patients treated with the combination of rituximab and chemotherapy in first line, which have been refractory or relapsed after having achieved any responses to this first line of pretreatment (excluding radiotherapy).
4. ECOG ≤ 2.
5. Signed written informed consent.

Exclusion Criteria:

1. Clinical suspicion or documentation of histological transformation.
2. Have received prior chemotherapy scheme, first line without Rituximab.
3. Prior autologous or allogeneic.
4. CNS infiltration by LF (primary CNS lymphoma or lymphomatous meningitis).
5. Past or active Hepatitis B (at least one of the following markers HBsAg, HBe Ag, anti-HBc, HBV DNA)
6. HCV infection. HIV infection or other conditions of serious immunosuppression.
7. Previous neoplasms except non-melanoma skin cancer of the cervix or adequately treated.
8. Cardiac function in cardiac patient known or prior treatment with anthracyclines with EF <50%.
9. Impaired renal function (creatinine> 1.5 x Upper Limit of Normal, LSN) or a creatinine clearance <50 ml / h, not related to lymphoma.
10. Impaired liver function (bilirubin, AST / ALT or GGT> 2 x ULN) were not related to lymphoma.
11. Women who are nursing or pregnant. Women of childbearing potential will be included prior pregnancy test serum / urine negative. Use effective contraception to be kept for 1 year after cessation of rituximab.
12. Patients with heart disease, pulmonary, neurological, psychiatric or severe metabolic and not secondary to lymphoma.
13. Severe acute or chronic infection in activity.
14. Any other concurrent medical or psychological comorbidity that might interfere with participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Peñalver Párraga, MD, Principal Investigator — Hospital Universitario Fundación Alcorcón; Javier De la Serna Torroba, MD, Principal Investigator — Hospital 12 de Octubre; Francisca Oña Compan, MD, Principal Investigator — Hospital de Getafe.; Patricia Font López, MD, Principal Investigator — Gregorio Marañón Hospital; Secundino Ferrer Bordas, MD, Principal Investigator — Hospital Dr. Peset; José Ramón Mayans Ferrer, MD, Principal Investigator — Hospital Arnau de Vilanova; Eulogio Conde García, MD, Principal Investigator — Hospital Marqués de Valdecilla; José Antonio Márquez Navarro, MD, Principal Investigator — Hospital de Basurto; Ernesto Pérez Persona, MD, Principal Investigator — Hospital Txagorritxu; Garazi Letamendi Madariaga, MD, Principal Investigator — Hospital de Galdakao; Pilar Giraldo Castellanos, MD, Principal Investigator — Hospital Miguel Servet; Luis Palomera Bernal, MD, Principal Investigator — Hospital Clínico de Zaragoza; Andrés López Hernández, MD, Principal Investigator — Hospital Vall d´Hebron; Blanca Sánchez González, MD, Principal Investigator — Hospital del Mar; José Luis Sánchez-Majado, MD, Principal Investigator — Hospital San Juan de Alicante; Antonio Gutiérrez García, MD, Principal Investigator — Hospital Son Espases; Francisco Javier Capote Huelva, MD, Principal Investigator — Hospital Universitario Puerta del Mar; Fátima de la Cruz, MD, Principal Investigator — Hospital Virgen del Rocío; Mª José Ramírez, MD, Principal Investigator — Hospital de Jerez; Fernando Carnicero González, MD, Principal Investigator — Hospital San Pedro de Alcantara; Mª José Rodríguez Salazar, MD, Principal Investigator — Hospital Universitario de Canarias; Miguel Ángel Canales Albendea, MD, Principal Investigator — Hospital La Paz; José Antonio García Marco, MD, Principal Investigator — Hospital Puerta de Hierro; Carlos Montalbán Sanz, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Rosalía Riaza Grau, MD, Principal Investigator — Hospital Severo Ochoa; Mª Dolores Caballero Barrigón, MD, Principal Investigator — Hospital de Salamanca; Mª Jesús Peñarrubia Ponce, MD, Principal Investigator — Hospital Río Hortega; José Antonio Queizán, MD, Principal Investigator — Hospital de Segovia; Roberto Hernández Martín, MD, Principal Investigator — Hospital Virgen de la Concha; Mª José Terol Castera, MD, Principal Investigator — Hospital Clínico de Valencia; Félix Carbonell, MD, Principal Investigator — Hospital General Universitario de Valencia; María Rosario Varela Gómez, MD, Principal Investigator — Complejo Hospitalario A Coruña; José Luis Bello López, MD, Principal Investigator — C. H. U. Santiago; Carlos Panizo, MD, Principal Investigator — Clínica Universitaria de Navarra; Juan Manuel Sancho Cia, MD, Principal Investigator — Germans Trias i Pujol Hospital; Armando López Guillermo, MD, Principal Investigator — Hospital Clínic i Provincial; Elena Pérez Ceballos, MD, Principal Investigator — Hospital Morales Meseguer; Andrés Sánchez Salinas, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca; Mª Soledad Durán Nieto, MD, Principal Investigator — Hospital de Jaén; Manuel Espeso de Haro, MD, Principal Investigator — Hospital Carlos Haya; Joan Bargay Lleonart, MD, Principal Investigator — Hospital Son Llàtzer
Locations (41):
- Spain (41):
  - Complejo Hospitalario Universitario de Santiago, Santiago, A Coruña
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital San Juan de Alicante, Sant Joan d'Alacant, Alicante
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Galdakao, Galdakao, Bilbao
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital de Getafe, Getafe, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Virgen de Arrixaca, El Palmar, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Puerta del Mar, Cadiz
  - Hospital San Pedro Alcántara, Cáceres
  - Hospital de Jaén, Jaén
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Complejo Hospitalario Carlos Haya, Málaga
  - Hospital Morales Meseguer, Murcia
  - Hospital de Salamanca, Salamanca
  - Hospital General de Segovia, Segovia
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Río Hortega, Valladolid
  - Hospital Virgen de la Concha, Zamora
  - Hospital Clínico de Zaragoza, Zaragoza
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Penalver FJ, Marquez JA, Duran S, Giraldo P, Martin A, Montalban C, Sancho JM, Ramirez MJ, Terol MJ, Capote FJ, Gutierrez A, Sanchez B, Lopez A, Salar A, Rodriguez-Caravaca G, Canales M, Caballero MD; GELTAMO (The Spanish Lymphoma Cooperative Group). Response-adapted treatment with rituximab, bendamustine, mitoxantrone, and dexamethasone followed by rituximab maintenance in patients with relapsed or refractory follicular lymphoma after first-line immunochemotherapy: Results of the RBMDGELTAMO08 phase II trial. Cancer Med. 2019 Nov;8(16):6955-6966. doi: 10.1002/cam4.2555. Epub 2019 Oct 1. PMID 31573746

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab, Bendamustine, Mitoxantrone, Dexamethasone: Patient will receive Rituximab, Bendamustina, Mitoxantrone and Dexametasona
  Rituximab, Bendamustine, Mitoxantrone, Dexamethasone: Bendamustine: 90 mg/m2/day, days 1 and 2 of each cycle, iv Mitoxantrone: 6 mg/m2/day, day 1 of each cycle, iv DEXAMETHASONE 20 mg / day, days 1 through 5 of each cycle, od Rituximab: 375 mg / m 2 / day, day 1 of each cycle, iv
Period: Overall Study
Arm/Group | Rituximab, Bendamustine, Mitoxantrone, Dexamethasone
Started | 60
Completed | 43
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab, Bendamustine, Mitoxantrone, Dexamethasone
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 28
Age, Continuous [Median (Full Range); unit: years] | 62 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30
Region of Enrollment [Number; unit: participants]
  Spain | 60

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The primary endpoint is the number of Participants with Response according to the criteria of the International Workshop to Standardize Response Criteria for NHL
  Complete Remission (CR):
  Nodes returned to normal (if GTD >15 mm before therapy, GTD now ≤15 mm; if GTD 11-15 and SA >10 mm before therapy, SA now ≤10 mm) All (non-nodal) target lesions completely resolved
  Partial Remission (PR) SPD of target lesions decreased ≥50% from baseline Spleen and liver nodules regress by 50% in SPD or single lesion in GTD
  Stable Disease (SD) Not enough shrinkage for PR Not enough growth for PD
  Progressive Disease (PD):
  SPD increase ≥50% from nadir (smallest value seen during trial) in nodal target lesions overall or in any single nodal target lesion
Time Frame: 7 years
Population: Number of Participants analyzed in the Maintenance Rituximab Arm reflects all participants who received at least one dose of Rituximab during maintenance, and had available data for response during that phase
Measure: Count of Participants; unit: Participants
Groups:
- Induction Rituximab, Bendamustine, Mitoxantrone, Dexamethasone: Patient will receive Rituximab, Bendamustina, Mitoxantrone and Dexametasona
  Rituximab, Bendamustine, Mitoxantrone, Dexamethasone: Bendamustine: 90 mg/m2/day, days 1 and 2 of each cycle, iv Mitoxantrone: 6 mg/m2/day, day 1 of each cycle, iv DEXAMETHASONE 20 mg / day, days 1 through 5 of each cycle, od Rituximab: 375 mg / m 2 / day, day 1 of each cycle, iv
- Maintenance Rituximab: Patient who had response to induction will receive Rituximab in maintenance
  Rituximab: 375 mg / m2 every three months
Arm/Group | Induction Rituximab, Bendamustine, Mitoxantrone, Dexamethasone | Maintenance Rituximab
Number analyzed (Participants) | 60 | 43
Participants | 57 | 35

2. Secondary Outcome: Secondary Endpoints Included an Assessment of the Following Parameters: Progression-Free Survival, Disease-Free Survival, Global Survival, Duration of the Response.
Time Frame: 7 years
Population: Only those patients who started the maintenance treatmet were analyzed for Disease-Free Survival
Measure: Median (Full Range); unit: months
Arm/Group | R-BMD
Number analyzed (Participants) | 60
months
  Progression-Free Survival | 56 [28 to 56]
  Disease-Free Survival: number analyzed (Participants) | 45
  Disease-Free Survival | 51 [36 to NA] — Insufficient number of participants with events. Superior data to Disease-Free Survival is still not available
  Global Survival | NA [NA to NA] — Insufficient number of participants with events. Global Survival data is still not available
  Duration of the Response | 54 [36 to 54]

ADVERSE EVENTS:
Time Frame: 9 years
Groups:
- Rituximab, Bendamustine, Mitoxantrone, Dexamethasone: Patient will receive Rituximab, Bendamustina, Mitoxantrone and Dexametasona
  Rituximab, Bendamustine, Mitoxantrone, Dexamethasone: Bendamustine: 90 mg/m2/day, days 1 and 2 of each cycle, iv Mitoxantrone: 6 mg/m2/day, day 1 of each cycle, iv DEXAMETHASONE 20 mg / day, days 1 through 5 of each cycle, od Rituximab: 375 mg / m 2 / day, day 1 of each cycle, iv
  Patients with response will receive Rituximab in maintenance: 375 mg / m2 every three months
Arm/Group | Rituximab, Bendamustine, Mitoxantrone, Dexamethasone
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 22/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab, Bendamustine, Mitoxantrone, Dexamethasone (N=60)
Infection (Infections and infestations) | 12 (20)
Diarrhea (Gastrointestinal disorders) | 2 (5)
Fever (General disorders) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (6)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Leucoencephalopathy (Nervous system disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (2)
Surgery (Surgical and medical procedures) | 3 (3)
Progression suspicion (Investigations) | 1 (1)
Oral ulcer (Gastrointestinal disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Arthritis (Immune system disorders) | 1 (2)
Hepatic insufficiency (Metabolism and nutrition disorders) | 1 (1)
Immunodeficiency (Metabolism and nutrition disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neuropathy caranial-CN VII (Nervous system disorders) | 1 (1)
Pleural effussion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab, Bendamustine, Mitoxantrone, Dexamethasone (N=60)
Neutropenia (Blood and lymphatic system disorders) | 50 (318)
Anemia (Blood and lymphatic system disorders) | 43 (144)
plateletes (Blood and lymphatic system disorders) | 41 (135)
pain (General disorders) | 21 (58)
Infection (Infections and infestations) | 40 (79)
fatigue (General disorders) | 18 (36)
Metabolic/laboratory (Metabolism and nutrition disorders) | 45 (82)
Fever (General disorders) | 20 (25)
Diarrhea (Gastrointestinal disorders) | 11 (21)
Vomiting (Gastrointestinal disorders) | 11 (15)
Allergic reaction (Immune system disorders) | 8 (11)
mucositis (Skin and subcutaneous tissue disorders) | 3 (11)
constipation (Gastrointestinal disorders) | 8 (10)
Febrile neutropenia (Infections and infestations) | 6 (6)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
cold (Respiratory, thoracic and mediastinal disorders) | 5 (8)
mood alteration (Psychiatric disorders) | 5 (7)
pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (5)
other (Blood and lymphatic system disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 4 (4)
hearing (Ear and labyrinth disorders) | 4 (7)
dispnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No